CLINICAL TRIAL: NCT06966141
Title: A Real World Study: Clinical Outcomes and Safety of Sacituzumab Govitecan in Metastatic HER-2 Negative Breast Cancer Patients
Brief Title: A Real World Study of Sacituzumab Govitecan
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Professor, Fudan University
Other Study IDs: WONDER
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Metastatic; Treatment Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients received SG: HER2-negative breast cancer patients who received SG in the advanced stage

SUMMARY:
Clinical Outcomes and Safety of Sacituzumab Govitecan in Metastatic HER-2 negative Breast Cancer Patients

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 or above;
2. The Eastern Cooperative Oncology Group (ECOG) physical condition score of the United States is ≤2;
3. Unresectable or metastatic triple-negative breast cancer confirmed by tumor histology or cytology, and having received at least two systemic treatments previously (at least one of which was for metastatic disease); Or HR+/HER2- (IHC 0, 1+ or IHC 2+/ISH-) unresectable or metastatic breast cancer confirmed by tumor histology or cytology, with previous endocrine therapy and ≥2 lines of systemic therapy (for metastatic disease);
4. Receive gosatetuzumab treatment in the advanced stage;
5. During the study period, voluntarily abide by this trial protocol and receive regular follow-ups;
6. All women of childbearing age, fertile men or their spouses who have no plans for fertility or sperm donation throughout the trial period until 6 months after the last dose, or who voluntarily take effective contraceptive measures.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Those with acute or chronic infections, or those with other serious diseases at the same time, are judged by the researchers as unsuitable for this study;
3. Having suffered from other malignant tumors within 5 years (excluding the following situations: cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary thyroid carcinoma; A second primary cancer that has been completely cured and has no recurrence within five years; Researchers have clearly identified which primary tumor source the metastatic foci belong to.
4. Those with mental illness or mental disorders, poor compliance and inability to cooperate and describe treatment responses;
5. Those with severe organic diseases or major organ failure, such as decompensated heart, lung, liver or kidney failure, which makes them unable to tolerate treatment;
6. Patients allergic to gosatetuzumab;
7. Patients who changed their treatment regimens after gosatetuzumab treatment due to non-disease progression reasons;
8. The researcher believes that the patient has other circumstances that make them unsuitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER-2 negative Breast Cancer Patients received SG
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
PFS | Six months after the last patient was enrolled
  PFS was defined as the time interval from the date of DS-8201 initiation until date of progressive disease (PD) or death from any causes, whichever occurred first.
ORR | Up to approximately 12 weeks
  ORR is the percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, MD,PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China